CLINICAL TRIAL: NCT04276558
Title: Efficacy, Safety and Pharmacokinetics of 3 Doses of REC 0/0559 Eye Drops for the Treatment of Stage 2 (Moderate) and 3 (Severe) Neurotrophic Keratitis in Adult Patients
Brief Title: REC 0/0559 Eye Drops for Treatment of Moderate and Severe Neurotrophic Keratitis in Adult Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RECORDATI GROUP (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: REC0559-B-001
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Neurotrophic Keratitis

STUDY DESIGN:
Intervention Model Description: The study will have an initial period of dose escalation followed by a parallel recruitment period. Randomisation in the first 24 patients will be sequential and after, patients will be randomised to all 4 treatment arms.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-masked: dose and nature of the product
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose 1 - 0.5 µg/day (Experimental): Dose of study drug per day: 0.5 µg/day Study drug concentration: 5 µg/mL MT8 given 1 drop QID
  Interventions: Drug: Udonitrectag; Other: Vehicle
- Dose 2 - 2.5 µg/day (Experimental): Dose of study drug per day: 2.5 µg/day Study drug concentration: 25 µg/mL MT8 given 1 drop QID
  Interventions: Drug: Udonitrectag; Other: Vehicle
- Dose 3 - 5 µg/day (Experimental): Dose of study drug per day: 5 µg/day Study drug concentration: 50 µg/mL MT8 given 1 drop QID
  Interventions: Drug: Udonitrectag; Other: Vehicle
- Vehicle (Placebo Comparator): Dose of study drug per day: 0 µg/day Study drug concentration: Vehicle given 1 drop QID
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: Udonitrectag — Eye drop solution in single dose unit.
  Other Names: REC 0/0559
  Arms: Dose 1 - 0.5 µg/day; Dose 2 - 2.5 µg/day; Dose 3 - 5 µg/day
Other: Vehicle — Eye drop solution with no active substance in single dose unit.

SUMMARY:
A phase 2 study, aiming to evaluate the efficacy, safety and pharmacokinetics of REC 0/0559 in treatment of Neurotrophic Keratitis in Adult Patient in Europe and United States of America.

DETAILED DESCRIPTION:
This was a Phase 2, international, multicentre, dose-ranging, double-masked, randomised, parallel-group, vehicle-controlled study designed to evaluate 3 different doses of REC 0/0559 vs vehicle in patients with Stage 2 and Stage 3 neurotrophic keratitis (NK).

ELIGIBILITY:
Inclusion Criteria:

1. Have read, understood, and signed the informed consent form (ICF).
2. Be a male or female aged ≥18 years at the time of ICF signature.
3. Have stage 2 moderate (PED) or stage 3 severe (corneal ulcer) NK involving only 1 eye (study eye) and of at least 2 weeks duration. Patients with Stage 1 NK in the fellow eye can be enrolled.

   for the study eye
4. Have no objective clinical evidence of improvement in the PED or corneal ulceration within the 2 weeks before the screening visit despite use of conventional non-surgical treatment (eg, nonpreserved ocular lubricants, nonpreserved topical antibiotics, oral doxycycline, patching, serum tears, and/or therapeutic contact lenses) as determined by the investigator's or referring physician's medical record.
5. Have decreased corneal sensitivity (≤ 4 cm using the Cochet-Bonnet aesthesiometer) within the area of the PED or corneal ulcer and outside of the area of the defect in at least one corneal quadrant.
6. Have a BCDVA score ≤ 75 ETDRS letters in the study eye, due to NK.

Exclusion Criteria:

1. Have participated in any clinical trial with an investigational drug/device within 2 months before the Screening Visit and throughout the study duration.
2. Have a known hypersensitivity to one of the components of the study drug or procedural medications (eg, fluorescein), including to a compound chemically related to MT8
3. Have a presence or history of any ocular or systemic disorder or condition that might hinder the efficacy of the study treatment or its evaluation, could possibly interfere with the interpretation of study results, or could be judged by the investigator to be incompatible with the study visit schedule or conduct (eg, progressive or degenerative corneal or retinal conditions, lagophthalmos, uveitis, optic neuritis, poorly controlled diabetes, autoimmune disease, systemic infection, neoplastic diseases), or that may compromise the safety of the patient.
4. Have a significant history of alcohol abuse or drug/solvent abuse
5. Be unwilling to comply with any study assessments or procedures.
6. Be a woman who is pregnant, nursing or planning a pregnancy.
7. Be a woman of childbearing potential not using a highly effective method of birth control.
8. Be a male patient who is not permanently sterile and who is not willing to use condoms during the study and for 4 weeks after the end of study treatment.

   For the study eye:
9. Have any active ocular infection (bacterial, viral, fungal or protozoal) or active inflammation not related to NK in the study eye.
10. Have any other ocular disease requiring topical ocular treatment in the study eye during the course of the study treatment period, except for glaucoma if treated by preservative-free eye drop (single-agent treatment, once daily, stable regimen 4 weeks before screening and during the study),
11. Receive topical ophthalmological treatments other than the study drug provided by the study Sponsor and the treatments allowed by the study protocol (eg, preservative-free artificial tears; preservative-free eye drop (single-agent treatment, once daily, stable regimen 4 weeks before screening and during the study) for glaucoma; topical antibiotics; other than tetracycline).
12. Have severe blepharitis and/or severe meibomian gland disease in the study eye.
13. Have severe vision loss in the study eye with no potential for visual improvement in the opinion of the investigator as a result of the study treatment.
14. Have evidence of corneal ulceration/melting involving the posterior third of the corneal stroma, or perforation in the study eye.
15. Have a history of any ocular surgery (including laser or refractive surgical procedures) within 3 months before the Screening Visit in the study eye. An exception to the preceding statement will be allowed if the ocular surgery is considered to be the cause of the Stage 2 or 3 NK.
16. Have a history of corneal transplantation in the study eye, except if performed to treat NK and at least 6 months prior screening.
17. Have had prior surgical procedures for the treatment of NK (eg, tarsorrhaphy, conjunctival flap, etc.) except AMT, if at least 2 wks after the membrane has disappeared within the area of the PED or corneal ulcer (and at least 6 weeks after the procedure) in the study eye.
18. Use therapeutic contact lenses or wear contact lenses for refractive correction during the study treatment periods in the eye(s) with NK.
19. Have an anticipated need for punctal occlusion during the study treatment period. Patients with punctal occlusion or punctal plugs inserted before the study are eligible for enrolment provided that the punctal occlusion is maintained during the study.
20. Have an uncontrolled glaucoma at the Screening Visit. (Patients suffering from glaucoma requiring ophthalmic drops for topical treatment at the Screening Visit or during the study are not eligible, except if the ophthalmic drops is a preservative-free treatment administered maximum once daily as a single-agent treatment and at a stable regimen 4 weeks before screening and at the same dose during the study. Patients treated with oral intraocular pressure-lowering drugs at the Screening Visit and during the study may be enrolled if their glaucoma status is assessed as stable and controlled.

    For the fellow eye
21. Have Stage 2 or 3 NK or perforation.

    For any eye:
22. Have a history of ocular cancer.
23. Have had prior treatment with Oxervate™

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (9):
  - Nature Coast Clinical Research, Crystal River, Florida
  - University of Florida, Gainesville, Florida
  - University of Maryland School of Medicine UMSOM, Baltimore, Maryland
  - University of Michigan - Kellogg Eye Center, Ann Arbor, Michigan
  - Mt. Sinai New York Eye and Ear Infirmary, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Toyos Clinic, Nashville, Tennessee
  - Houston Eye Associates HEA - Gramercy Location, Houston, Texas
  - University of Wisconsin-Madison, Madison, Wisconsin
- France (4):
  - Dijon University Hospital CHU Dijon, Dijon
  - CHU Paris Centre - Hôpital Cochin, Paris
  - Hôpital Fondation Adolphe de Rothschild, Paris
  - Hôpital Universitaire Necker, Paris
- Germany (6):
  - Ludwig-Maximilians-Universitaet Muenchen LMU - Augenklinik, Munich, Bavaria
  - Uniklinik Koeln, Cologne
  - Hospital Eye University of Duesseldorf, Düsseldorf
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Saarland University Medical Center, Homburg
  - UNIVERSITÄTSMEDIZIN der Johannes Gutenberg-Universität Mainz, Mainz
- Hungary (3):
  - Markusovszky University Teaching Hospital, Szombathely, Vas County
  - Semmelweis University, Dept. of Ophthalmology, Budapest
  - University of Pecs - Dpt of Ophthalmology, Pécs
- Italy (9):
  - Università Magna Grecia di Catanzaro, Germaneto, Calabria
  - Azienda Universitaria Ospedaliera Consorziale - Policlinico Bari Clinica Oculistica, Bari
  - DIMES Universit di Bologna, Bologna
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedali Privato, Forlì
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Azienda Ospedaliera Universitaria Policlinico Gaetano Martino, Messina
  - Ospedale Luigi Sacco, Milan
  - Fondazione PTV - Policlinico Tor Vergata, Roma
- Spain (6):
  - Instituto Oftalmologico Fernandez-Vega, Oviedo, Principality of Asturias
  - Hospital de Cruces, Barakaldo
  - Instituto Microcirugia Ocular IMO, Barcelona
  - Centro de Oftalmologia Barraquer, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Cartuja Vision - Centro de Servicios Oftlamologicos, Seville
- United Kingdom (4):
  - Royal Liverpool University Hospital - St Paul's Clinical Eye Research Centre, Liverpool, Mersey
  - University Hospital Hairmyres, Glasgow
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 108 patients were randomised, and all of them received at least one dose of study drug. A total of 83 patients (76.9%) completed the 8-week treatment period and 88 patients (81.5%) completed the study regardless of the study treatment duration. The drug was instilled in 1 study eye per participant.
Units Other Than Participants: eye
Period: Overall Study
Arm/Group | Dose 1 - 0.5 µg/Day | Dose 2 - 2.5 µg/Day | Dose 3 - 5 µg/Day | Vehicle
Started | 27; 27 eye | 26; 26 eye | 26; 26 eye | 29; 29 eye
Completed | 23; 23 eye | 21; 21 eye | 21; 21 eye | 23; 23 eye
Not Completed | 4; 4 eye | 5; 5 eye | 5; 5 eye | 6; 6 eye

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose 1 - 0.5 µg/Day | Dose 2 - 2.5 µg/Day | Dose 3 - 5 µg/Day | Vehicle | Total
Number analyzed (Participants) | 27 | 26 | 26 | 29 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (14.05) | 59.6 (15.30) | 65.6 (17.14) | 67.0 (16.76) | 65.7 (16.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 14 | 14 | 52
  Male | 14 | 15 | 12 | 15 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 4 | 4 | 5 | 16
  Unknown or Not Reported | 24 | 22 | 22 | 23 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 0 | 3
  White | 26 | 21 | 19 | 27 | 93
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 4 | 4 | 2 | 11
Region of Enrollment [Number; unit: participants]
  Hungary | 1 | 1 | 0 | 3 | 5
  United States | 3 | 4 | 4 | 6 | 17
  Italy | 13 | 6 | 6 | 7 | 32
  United Kingdom | 2 | 2 | 3 | 3 | 10
  France | 1 | 1 | 2 | 2 | 6
  Germany | 6 | 10 | 9 | 4 | 29
  Spain | 1 | 2 | 2 | 4 | 9
Height [Mean (Standard Deviation); unit: cm] | 166.694 (9.5229) | 171.99 (9.5848) | 169.598 (12.1409) | 167.662 (14.8453) | 168.748 (11.7409)
Weight [Mean (Standard Deviation); unit: kg] | 79.051 (19.1023) | 77.379 (22.5637) | 72.377 (14.5292) | 74.718 (19.6181) | 75.889 (19.0756)

OUTCOME MEASURES:

1. Primary Outcome: Corneal Healing
Description: The primary endpoint of this study is the percentage of patients achieving complete corneal healing of PED or corneal ulcer at Week 8, defined as no corneal fluorescein staining in the area of the PED or corneal ulcer as assessed by an independent central reading centre.
Time Frame: At week 8
Population: The total patients were divided in subgroups according to disease stage (moderate or severe) and Region (EU or NA)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 - 0.5 µg/Day | Dose 2 - 2.5 µg/Day | Dose 3 - 5 µg/Day | Vehicle
Number analyzed (Participants) | 27 | 26 | 26 | 29
Participants
  Disease stage 2 (moderate) EU: number analyzed (Participants) | 10 | 11 | 10 | 11
  Disease stage 2 (moderate) EU: Healed | 4 | 2 | 1 | 2
  Disease stage 2 (moderate) EU: Not healed | 6 | 9 | 9 | 9
  Disease stage 3 (Severe) EU: number analyzed (Participants) | 14 | 11 | 12 | 12
  Disease stage 3 (Severe) EU: Healed | 3 | 2 | 3 | 5
  Disease stage 3 (Severe) EU: Not healed | 11 | 9 | 9 | 7
  Disease stage 2 (moderate) NA: number analyzed (Participants) | 2 | 2 | 2 | 3
  Disease stage 2 (moderate) NA: Healed | 2 | 0 | 0 | 0
  Disease stage 2 (moderate) NA: Not healed | 0 | 2 | 2 | 3
  Disease stage 3 (Severe) NA: number analyzed (Participants) | 1 | 2 | 2 | 3
  Disease stage 3 (Severe) NA: Healed | 0 | 1 | 1 | 3
  Disease stage 3 (Severe) NA: Not healed | 1 | 1 | 1 | 0

2. Secondary Outcome: Visual Acuity
Description: Percentage of patients who achieve a 5-, 10-, and 15-letter mean improvement in best corrected distance visual acuity (BCDVA) by Early Treatment Diabetic Retinopathy Study (ETDRS) chart at Week 8 compared to baseline (in all patients and in patients with a central location of the PED or corneal ulcer, respectively).
Time Frame: At week 8
Population: The population was analysed in subgroups according to the location of the PED or corneal ulcer (central versus all locations).
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 - 0.5 µg/Day | Dose 2 - 2.5 µg/Day | Dose 3 - 5 µg/Day | Vehicle
Number analyzed (Participants) | 27 | 26 | 26 | 29
Participants
  Improvement ≥ 5 letters (all locations): Improved | 9 | 11 | 10 | 7
  Improvement ≥ 5 letters (all locations): Not improved | 18 | 15 | 16 | 22
  Improvement ≥ 10 letters (all locations): Improved | 7 | 9 | 6 | 6
  Improvement ≥ 10 letters (all locations): Not improved | 20 | 17 | 20 | 23
  Improvement ≥ 15 letters (all locations): Improved | 7 | 5 | 5 | 6
  Improvement ≥ 15 letters (all locations): Not improved | 20 | 21 | 21 | 23
  Improvement ≥ 5 letters (central PED or central corneal ulcer): number analyzed (Participants) | 21 | 24 | 19 | 19
  Improvement ≥ 5 letters (central PED or central corneal ulcer): Improved | 4 | 10 | 7 | 5
  Improvement ≥ 5 letters (central PED or central corneal ulcer): Not improved | 17 | 14 | 12 | 14
  Improvement ≥ 10 letters (central PED or central corneal ulcer): number analyzed (Participants) | 21 | 24 | 19 | 19
  Improvement ≥ 10 letters (central PED or central corneal ulcer): Improved | 3 | 8 | 5 | 4
  Improvement ≥ 10 letters (central PED or central corneal ulcer): Not improved | 18 | 16 | 14 | 15
  Improvement ≥ 15 letters (central PED or central corneal ulcer): number analyzed (Participants) | 21 | 24 | 19 | 19
  Improvement ≥ 15 letters (central PED or central corneal ulcer): Improved | 3 | 5 | 4 | 4
  Improvement ≥ 15 letters (central PED or central corneal ulcer): Not improved | 18 | 19 | 15 | 15

ADVERSE EVENTS:
Time Frame: Safety assessments were conducted for all patients from the Screening Visit (upon the signature of the ICF) to the end of the study (8 weeks)
Arm/Group | Dose 1 - 0.5 µg/Day | Dose 2 - 2.5 µg/Day | Dose 3 - 5 µg/Day | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/27 | 1/26 | 0/26 | 0/29
Serious Adverse Events (participants affected / at risk) | 4/27 | 3/26 | 7/26 | 4/29
Other Adverse Events (participants affected / at risk) | 18/27 | 17/26 | 18/26 | 11/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose 1 - 0.5 µg/Day (N=27) | Dose 2 - 2.5 µg/Day (N=26) | Dose 3 - 5 µg/Day (N=26) | Vehicle (N=29)
Ulcerative keratitis (Eye disorders) | 1 | 1 | 3 | 1 — in study eye
Corneal epithelium defect (Eye disorders) | 1 | 0 | 0 | 0 — in study eye
Corneal erosion (Eye disorders) | 0 | 1 | 0 | 0 — study eye
Corneal perforation (Eye disorders) | 0 | 0 | 1 | 0 — in study eye
Sudden visual loss (Eye disorders) | 0 | 0 | 0 | 1 — in study eye
Herpes ophthalmic (Infections and infestations) | 0 | 0 | 1 | 0 — in study eye
Hypopyon (Infections and infestations) | 0 | 0 | 1 | 0 — in study eye
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 — in study eye
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Coronavirus infection (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Wound sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Corneal graft rejection (Immune system disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3.7% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose 1 - 0.5 µg/Day (N=27) | Dose 2 - 2.5 µg/Day (N=26) | Dose 3 - 5 µg/Day (N=26) | Vehicle (N=29)
Neutrophic keratopathy (Eye disorders) | 2 | 2 | 3 | 4 — in study eye
Eye pain (Eye disorders) | 1 | 5 | 1 | 3 — in 1 fellow eye for vehicle and study eyes for the rest of participants
Ulcerative keratitis (Eye disorders) | 1 | 1 | 3 | 3 — in study eye
Visual acuity reduced (Eye disorders) | 0 | 3 | 3 | 3 — in study eye
Conjunctival hyperemia (Eye disorders) | 2 | 1 | 0 | 1 — in study eye
Corneal oedema (Eye disorders) | 0 | 4 | 0 | 0 — 1 in fellow eye and 3 in study eyes
Eye irritation (Eye disorders) | 0 | 2 | 2 | 0 — in study eye
Eye pruritus (Eye disorders) | 0 | 1 | 2 | 1 — in study eye
Corneal scar (Eye disorders) | 0 | 2 | 0 | 1 — in study eye
Foreign body sensation in eyes (Eye disorders) | 0 | 2 | 1 | 0 — in study eye
Hypoaesthesia eye (Eye disorders) | 0 | 2 | 0 | 1 — in study eye
Corneal opacity (Eye disorders) | 0 | 2 | 0 | 0 — in study eye
Lacrimation increased (Eye disorders) | 1 | 2 | 0 | 0 — in study eye
Visual impairment (Eye disorders) | 0 | 2 | 0 | 0 — in study eye
Coronavirus infection (Infections and infestations) | 1 | 3 | 3 | 0
Influenza (Infections and infestations) | 0 | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 0
Corneal epithelium defect (Eye disorders) | 2 | 2 | 2 | 1 — in study eye
Corneal erosion (Eye disorders) | 1 | 1 | 0 | 0 — in fellow eye for dose 2, the rest in study eye
Corneal Perforation (Eye disorders) | 0 | 0 | 1 | 1 — in study eye
Crystoid macular oedema (Eye disorders) | 1 | 0 | 1 | 0 — in study eye for dose 1; fellow eye for dose 3
Ocular discomfort (Eye disorders) | 1 | 1 | 0 | 0 — in study eye
Ocular hyperemia (Eye disorders) | 0 | 1 | 1 | 0 — in study eye
Photophobia (Eye disorders) | 0 | 0 | 1 | 1 — in study eye
Vision Blurred (Eye disorders) | 0 | 1 | 0 | 1 — in study eye for vehicle and study eye for dose 2
Vitreous detachment (Eye disorders) | 1 | 0 | 0 | 1 — in study eye
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0 | 1 — in study eye
Abnormal sensation in the eye (Eye disorders) | 0 | 0 | 1 | 0 — in study eye
Anterior chamber flare (Eye disorders) | 0 | 1 | 0 | 0 — in study eye
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 — in fellow eye
Corneal deposits (Eye disorders) | 0 | 0 | 1 | 0 — in study eye
Corneal endothelitis (Eye disorders) | 0 | 1 | 0 | 0 — in study eye
Corneal neovascularisation (Eye disorders) | 0 | 0 | 1 | 0 — in study eye
Dellen (Eye disorders) | 0 | 1 | 0 | 0 — in study eye
Erythem of the eyelid (Eye disorders) | 0 | 1 | 0 | 0 — in study eye
Eye discharge (Eye disorders) | 0 | 1 | 0 | 0 — in study eye
Eyelids pruritus (Eye disorders) | 0 | 1 | 0 | 0 — in study eye
Keratitis (Eye disorders) | 0 | 1 | 0 | 0 — in study eye
Ocular surface disease (Eye disorders) | 0 | 1 | 0 | 0 — in study eye
Punctate keratitis (Eye disorders) | 0 | 0 | 1 | 0 — in study eye
Symblepharon (Eye disorders) | 1 | 0 | 0 | 0 — in study eye
Corneal infection (Infections and infestations) | 1 | 0 | 1 | 0 — in study eye
Hypopyon (Infections and infestations) | 0 | 1 | 1 | 0 — in study eye
Pneumonia (Eye disorders) | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Infective corneal ulcer (Infections and infestations) | 1 | 0 | 0 | 0 — in study eye
Keratitis bacterial (Eye disorders) | 1 | 0 | 0 | 0 — in study eye
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 — in study eye
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Wound sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 1 | 0
Blood tryglycerides increased (Investigations) | 1 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 1 | 0
lymphocytes count decreased (Investigations) | 0 | 1 | 0 | 1
White blood cell count increased (Investigations) | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood calcium increased (Investigations) | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0
Monocyte count increased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Instillation site irritation (General disorders) | 0 | 0 | 1 | 0 — in study eye
instillation site pain (General disorders) | 0 | 0 | 1 | 0 — in study eye
Instillation site pruritus (General disorders) | 0 | 0 | 1 | 0 — in study eye
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — in study eye
Corneal graft rejection (Immune system disorders) | 0 | 1 | 1 | 1 — in study eye
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure cogestive (Cardiac disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT04276558/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT04276558/SAP_001.pdf
  • Informed Consent Form (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT04276558/ICF_002.pdf